CLINICAL TRIAL: NCT03763981
Title: Comparison of Prolene Thread Seton Vs Silk Thread Seton for the Treatment of Perianal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, principal investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s5
Record Dates: First submitted 2018-07-10; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Perianal Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolene seton (Active Comparator): Prolene thread will be used as seton treatment for perianal fistulas
  Interventions: Procedure: prolene seton treatment
- silk seton (Active Comparator): Silk thread will be used as seton treatment for perianal fistulas
  Interventions: Procedure: silk seton treatment

INTERVENTIONS:
Procedure: prolene seton treatment — patients with perianal fistulas will treated with seton placement by prolene thread
  Arms: prolene seton
Procedure: silk seton treatment — patients with perianal fistulas will treated with seton placement by silk thread
  Arms: silk seton

SUMMARY:
It is a randomized control trial in which we will treat the patients with perianal fistula with seton placement. We will divide the patients in two groups. Group I will be treated with silk seton and Group II will be treated with prolene setone. The outcome will be then followed as fistula healing and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and aged 20 years and above with high perianal fistula

Exclusion Criteria:

* Low perianal fistulas Fistulas due to chrons disease, TB or carcinoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
fistula healing | 8 to 12 weeks
  fistula healing, complete healing of wound with no external opening of fistula

SECONDARY OUTCOMES:
Fistula recurrence | 6 months
  Recurrence of perianal fistula after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided